CLINICAL TRIAL: NCT03728179
Title: RACIN, A Phase I Study of the Combination of Nivolumab Associated With Low-dose Radiation, Aspirin/ Celecoxib, and Either Ipilimumab or Low-dose Cyclophosphamide, Followed by Nivolumab Maintenance, in Patients With Advanced, TIL-negative Solid Tumors
Brief Title: RACIN in Patients With Advanced TIL-negative Solid Tumors
Acronym: RACIN
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Dr Fernanda Herrera, Principal Investigator, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CHUV-DO-0003-RACIN_2017
Record Dates: First submitted 2018-10-15; First posted 2018-11-01 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Solid Tumor, Adult
MeSH Terms: interventions — Radiation; Nivolumab; Ipilimumab; Cyclophosphamide; Aspirin; Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Cohort 1 (Experimental): 0,5 Gy of RT + Cyclophosphamide + Nivolumab + Ipilimumab + Aspirin
  Interventions: Combination Product: Low dose irradiation + Nivolumab + Ipilimumab or Cyclophosphamide + Aspirin/Celecoxib
- Cohort 2 (Experimental): 1 Gy of RT + Cyclophosphamide + Nivolumab + Ipilimumab + Aspirin
  Interventions: Combination Product: Low dose irradiation + Nivolumab + Ipilimumab or Cyclophosphamide + Aspirin/Celecoxib
- Cohort 3a (Experimental): 1 Gy of RT + Cyclophosphamide + Nivolumab + Celecoxib
  Interventions: Combination Product: Low dose irradiation + Nivolumab + Ipilimumab or Cyclophosphamide + Aspirin/Celecoxib
- Cohort 4a (Experimental): 2 Gy of RT + Cyclophosphamide + Nivolumab + Celecoxib
  Interventions: Combination Product: Low dose irradiation + Nivolumab + Ipilimumab or Cyclophosphamide + Aspirin/Celecoxib
- Phase I b (Experimental): Recommended Phase Ib RT dose (RP1bD) + Nivolumab + Ipilimumab or Cyclophosphamide + Celecoxib
  Interventions: Combination Product: Low dose irradiation + Nivolumab + Ipilimumab or Cyclophosphamide + Aspirin/Celecoxib
- Cohort 3b (Experimental): 1 Gy of RT + Ipilimumab + Nivolumab + Celecoxib
  Interventions: Combination Product: Low dose irradiation + Nivolumab + Ipilimumab or Cyclophosphamide + Aspirin/Celecoxib
- Cohort 4b (Experimental): 2 Gy of RT + Ipilimumab + Nivolumab + Celecoxib
  Interventions: Combination Product: Low dose irradiation + Nivolumab + Ipilimumab or Cyclophosphamide + Aspirin/Celecoxib

INTERVENTIONS:
Combination Product: Low dose irradiation + Nivolumab + Ipilimumab or Cyclophosphamide + Aspirin/Celecoxib — Low Dose Radiation (RT): RT will be administered as single fractions every 2 weeks (Q2W) from cycle C0 to cycle C4. RT will be delivered to a number of metastatic deposits visible by PET/CT, at the PI's discretion.
  Cyclophosphamide: 200mg/m2 will be administered as intravenous infusion (IV) Q2W from cycle C0 to C4.
  Nivolumab: 240 mg will be administered as IV Q2W from cycle C1 to C4.
  Ipilimumab: 1mg/kg will be administered as IV every 6 weeks (Q6W) from cycle C1 to C4
  Aspirin: 300mg will be administered orally daily from cycle C1 to C4. All subjects will receive mandatory gastric prophylaxis with an oral H2 antagonist.
  Celecoxib: 200mg will be administered orally twice a day from cycle C1 to C4.
  At the end of cycle C4, patients eligible for maintenance will be treated with nivolumab at 240mg Q2W until progression or excessive toxicity; celecoxib will be maintained if the drug is well tolerated

SUMMARY:
Subjects with locally advanced or metastatic incurable Tumor Infiltrating Lymphocytes (TIL)-negative solid tumors who are not eligible for, declined or failed standard therapy will be treated with a combination nivolumab, low-dose ionizing radiation (RT) (0.5-2 Gy), aspirin (ASA)(cohorts 1 and 2)/celecoxib (cohorts 3, 4 and Phase Ib), and either ipilimumab or low-dose cyclophosphamide. The study comprises 2 phases: The aim of Phase Ia, is to determine safety and tolerability of a given combination therapy, as well as the maximum tolerated dose (MTD) or recommended phase Ib dose (RP1bD) of radiotherapy. Phase Ib aims to further explore safety and tolerability of this treatment in an expansion cohort.

In Phase Ia, 4 distinct cohorts will receive the following combination therapy:

Cohort1: combination therapy for 5 cycles (C0-C4) which includes: RT 0.5 Gy every 2 weeks (Q2W), Cy (200 mg/m2) Q2W (cycles C0 to C4); ASA (300 mg) daily, with nivolumab 240 mg flat dose Q2W and ipilimumab 1 mg/kg every 6 weeks (Q6W) will be administered (cycles C1 to C4).

Cohort2: combination therapy for 5 cycles (C0-C4) which includes: RT 1 Gy every 2 weeks (Q2W), Cy (200 mg/m2) Q2W (cycles C0 to C4); ASA (300 mg) daily, with nivolumab 240 mg flat dose Q2W and ipilimumab 1 mg/kg (Q6W) will be administered (cycles C1 to C4).

Cohorts 3a and 4a: Patients will receive Cy (200 mg/m2) Q2W, celecoxib (2x200mg daily), nivolumab (240 mg flat dose) Q2W, and low-dose radiation. Cohort 3a will receive 1 Gy of low-radiation dose and cohort 4a will receive 2 Gy.

Cohorts 3b and 4b: Patients will receive nivolumab (240 mg flat dose) Q2W, ipilimumab 1 mg/kg (Q6W), celecoxib (2x200mg daily) and low-dose radiation. Cohort 3b will receive 1 Gy of low-radiation dose and cohort 4b will receive 2 Gy.

In Phase Ia, the safety of combination (nivolumab, celecoxib, low-dose irradiation and cyclophosphamide) or (nivolumab, celecoxib, low-dose irradiation and ipilimumab) will be evaluated , and MTD or RP1bD will be defined. RP1bD will be the MTD or, in the absence of dose limiting toxicities (DLTs), the biologically best RT dose based on pharmacodynamics parameters.

In Phase Ib, patients will be treated with the MTD or RP1bD dose of RT and will follow the selected schema of treatment used in the Phase Ia cohort 3 or 4. At the end of the 5th cycle, patients eligible for nivolumab maintenance, will be treated with nivolumab at 240 mg Q2W until progression or excessive toxicity; celecoxib will be maintained according to tolerability.

ELIGIBILITY:
Pre-screening registration

Inclusion Criteria:

1. Signed pre-screening Informed Consent Form
2. Patients with recurrent or metastatic solid tumor (any histology), who progress after at least one standard therapy for advanced disease
3. Patient willingness and acceptance to participate in the immunology research is mandatory
4. At least one lesion accessible to biopsy without putting patient at risk
5. Biopsies obtained previously (within a maximum of 12 weeks before pre-screening visit), outside this protocol, for TIL assessment can be also considered for patient selection. Fresh tumor biopsies for subsequent translational studies will be used as baseline and collected at pre-screening (when biopsy will be performed for TIL status) or at screening (when archival biopsy will be used for TIL status). Biopsy from metastatic lymph nodes is accepted.
6. Eastern Cooperative Oncology Group (ECOG) clinical performance status: 0-1 for all patients, independently of the number of previous lines of therapy.
7. Life expectancy of ≥ 12 weeks
8. Patients with Glycose-6-Phosphate Dehydrogenase (G6PD) deficiency or any other hereditary coagulation disorder are excluded, as well as patients with clinical history of Reye syndrome
9. Adequate serology defined by the following laboratory results obtained during pre-screening period (day-28 to day-14).

   1. Seronegative for HIV infection (anti-HIV-1/-2)
   2. Seronegative for hepatitis B infection (HBs Ag, total anti-hemoglobin C (HBc), anti-HBs). Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen HBsAg test and a positive anti-HBc antibody test) are eligible, if hepatitis B virus (HBV) DNA test is negative.
   3. Seronegative for hepatitis C infection (anti-HCV): if a patient has positive anti-HCV antibody, a negative hepatitis C virus (HCV) RNA need to be obtain to register the patient.

Study registration

Inclusion Criteria

1. Signed main study Informed Consent Form
2. Absence of tumor-infiltrating intraepithelial Cluster of differentiation-8 positive T cells (CD8+ T cells) by immunohistochemistry (IHC) on baseline biopsy defined as <5 CD8+ cells per high power field of tumor
3. At least one lesion accessible to biopsy without putting patient at risk
4. Number of metastatic lesions viewed on Positron emission tomography-computed tomography (PET/CT) scan: for both Phase Ia and Phase Ib, the patient may have any number of metastatic lesions. A maximum of 10 metastatic lesions visible by PET/CT scan will be irradiated at the investigator's discretion. It is at the discretion of the investigator to exclude a metastatic site from the radiation field that, due to the radiotherapy volume, dose or location too close to a healthy organ, may put the patient at risk of suffering from radiation induced toxicity. If this would be the only metastatic site to be irradiated, the concerned patient will be excluded from the study.
5. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol
6. Adequate hematologic and end-organ function, defined by the following laboratory results obtained within 14 days prior to the first study treatment:

   1. Absolute neutrophil count ≥ 1.5 g/L (without granulocyte colony-stimulating factor support within 2 weeks prior registration)
   2. White Blood Cell (WBC) counts > 2.5 g/L and < 15 g/L
   3. Lymphocyte count ≥ 0.5 g/L
   4. Platelet count ≥ 100 g/L (without transfusion within 1 week prior registration)
   5. Hemoglobin ≥ 90 g/L (Patients may be transfused to meet this criterion but it should not be done within 1 week prior registration)
   6. Serum alanine aminotransferase (ALT), aspartate aminotransferase (AST) and alkaline phosphatase ≤ 2.5 x ULN (with the exception for patients with documented liver metastases: AST, ALT and alkaline phosphatase ≤ 5 x ULN)
   7. Serum bilirubin ≤ 1.5 x ULN (with the exception for: patients with known or suspicion of Gilbert disease who have serum bilirubin level ≤ 3 x ULN may be enrolled)
   8. Coagulation: International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or Partial Thromboplastin Time (PTT) is within therapeutic range of intended use of anticoagulants; Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
   9. Serum albumin > 25 g/L
   10. Serum creatinine ≤1.5 x ULN or creatinine clearance ≥ 40 ml/min on the basis of Cockcroft-Gault Formula
7. No prior radiation therapy in areas of desired radiation
8. Patients may have had prior therapy provided a washout period of 4 weeks prior to registration is allowed. Exception: hormone therapy for breast and prostate cancer is allowed to be continued during the study.
9. Recovery from any toxic effects of prior therapy before registration to ≤ Grade 1 per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v4.03) except for toxicities described below, as they do not put at risk the patient's condition and do not require systemic immunosuppressive steroids at any dose, including but not limited to: fatigue, alopecia, skin disorders, stable neuropathy, endocrinopathies requiring replacement treament.

   Note: for other medical conditions, or for any other toxicity with a higher grade but controlled by adequate treatment, prior discussion and agreement with the trial chair is mandatory.

   Note: Patients may have undergone surgical procedures within the past 3 weeks, as long as all toxicities have recovered to grade 1 or less.
10. For women of childbearing potential (WOCBP: sexually mature women who have not undergone a hysterectomy, have not been naturally post-menopausal for at least 12 consecutive months or have a serum follicle-stimulating hormone (FSH) < 40 Millions International Units (mIU)/ml):

    1. Agreement to use 2 acceptable methods of contraception during participation in the trial and for 6 months after last study combined treatment and after 5 months of maintenance treatment
    2. Women must have a negative urine pregnancy test within 7 days before registration. A positive urine test must be confirmed by a serum pregnancy test, or menopausal as per National Comprehensive Cancer Network (NCCN) guidelines.
11. For men: agreement to use 2 acceptable methods of effective contraception during participation in the trial and for 7 months after last study treatment (combined or maintenance treatment). Female partners of men who take part in this trial must also use at least one method of effective contraception during the trial and 7 months after last study treatment (combined or maintenance).

Exclusion Criteria:

1. Patients with soft tissue sarcoma, glioblastoma, or lymphoma are excluded.
2. Pregnant or breast-feeding women.
3. Symptomatic brain or leptomeningeal disease; any brain metastases must be stable for at least 6 months
4. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently)
5. Uncontrolled hypercalcemia (> 1.5 mmol/L ionized calcium or Ca > 12 mg/dL or corrected serum calcium > ULN) or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy or denosumab

   a) Patients who are receiving bisphosphonate therapy or denosumab specifically to prevent skeletal events and who do not have a history of clinically significant hypercalcemia are eligible.
6. Life expectancy of < 12 weeks
7. Current, recent (within 4 weeks prior to registration), or planned participation in an experimental drug study
8. New York Heart Association Class II or greater congestive heart failure
9. History of myocardial infarction or unstable angina within 6 months prior registration
10. History of stroke or transient ischemic attack within 6 months prior registration
11. Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior registration)
12. Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
13. Patients with active peptic or duodenal ulceration (within 4 weeks prior to registration)
14. Current or recent (within 14 days prior registration) treatment use of dipyramidole, ticlopidine, clopidogrel, cilostazol, prasugrel, or ticagrelor
15. Current or recent (within 14 days prior registration) use of full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic (as opposed to prophylactic) purpose

    1. Prophylactic anticoagulation for the patency of venous access devices is allowed, provided the activity of the agent results in an International Normalized Ratio (INR) < 1.5 x ULN and aPTT is within normal limits within 2 weeks prior registration.
    2. Prophylactic use of low molecular-weight heparin (e.g., enoxaparin) is allowed.
16. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins or allergy to biopharmaceuticals produced in Chinese hamster ovary cells
17. Known hypersensitivity to any component of the Investigational Medicinal Products (IMPs)
18. History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. The following exceptions are considered:

    1. Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone are eligible for this study.
    2. Patients with controlled Type I diabetes mellitus on a stable insulin regimen are eligible
19. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), druginduced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest Computerized Tomography (CT) scan. Exception: history of radiation pneumonitis in previous radiation field (fibrosis) is permitted provided that this area does not undergo current low dose irradiation as part of this protocol.
20. Severe infections within 4 weeks prior registration including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
21. Signs or symptoms of infection within 2 weeks prior registration
22. Received therapeutic oral or IV antibiotics within 2 weeks prior registration. Exception: patients receiving routine antibiotic prophylaxis (e.g., to prevent chronic obstructive pulmonary disease exacerbation or for dental extraction) are eligible.
23. Prior allogeneic stem cell or solid organ transplant
24. Administration of a live, attenuated vaccine within 4 weeks before registration. Exception: influenza vaccination should be given during influenza season only (approximately October to March). Patients must not receive live, attenuated influenza vaccine within 4 weeks prior registration or at any time during the study.
25. Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
26. Patients who have received prior treatment with anti-Programmed Cell Death-1 (PD1), anti-Programmed Cell Death Ligand-1 (PD-L1) or anti-Cytotoxic T-lymphocyte Associated 4 (CTLA-4) may be enrolled, provided at least 5 half-lives (approximately 75 days) have elapsed from the last dose to the registration and there was no history of severe immune-mediated adverse effects from such therapy (NCI CTCAE Grade 3 and 4).
27. Treatment with systemic immunostimulatory agents (including but not limited to interferon-alpha (IFN-a), interleukin-2 (IL-2)) for any reason within 6 weeks or five half-lives of the drug, whichever is shorter, prior registration
28. Treatment with systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor (anti-TNF) agents) within 2 weeks prior registration

    1. Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) or physiologic replacement doses (i.e., prednisone 5-7.5 mg/day) for adrenal insufficiency may be enrolled in the study.
    2. The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
Phases Ia and Ib: Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 3.5 years
  Phase Ia and IB: Toxicity and tolerability will be assessed through measure and evaluation of adverse events occuring during the study, using the National Cancer Institute (NCI) CommonTerminology Criteria for Adverse Events (CTCAE v.4.03)
Maximum Tolerated dose (MTD) or recommended phase Ib dose of low-dose irradiation for radio-immunotherapy combination (RP1bD). | 3.5 years
  MTD is defined as the dose level below the dose that causes a dose limiting toxicity (DLT) in more than 17% of participants. The MTD analysis population will consist of all evaluable participants registered in the phase Ia , who completed the DLT/ backbone limiting toxicity (BLT) period (cycle C0 and C1), unless discontinued due to toxicity. RP1bD will be the MTD or, in the absence of DLTs, the biologically best radiotherapy dose based on pharmacodynamics parameters.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 3.5 years
  Best objective response rate (Complete Response or Partial Response) during the period from enrolment to termination of trial treatment, will be assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1 or PCWG3 criteria for prostate cancer.
Disease Control Rate (DCR) | 6,12 and 24 months
  Percentage of patients achieving Complete Response, Partial Response or Stable Disease at the end of four cycles of combination therapy (i.e. at 6 months) as well as at 12 and 24 months, will be measured by RECIST v.1.1 or PCWG3 criteria for prostate cancer.
Progression free survival (PFS) rate | 6,12 and 24 months
  The time from enrolment until objective tumor progression or death, whichever occurs first, will be evaluated at 6,12 and 24 months by RECIST v.1.1 or PCWG3 criteria for prostate cancer.
Time to Progression (TTP): | 3.5 years
  The time from enrolment until objective tumor progression, will be evaluated by RECIST v.1.1 or PCWG3 criteria for prostate cancer.
Overall survival (OS) | 12 and 24 months
  OS will be assessed at 12 and 24 months

OTHER OUTCOMES:
Exploratory outcomes: Assessment of treatment response | 5 years
  Assessment of treatment response will be performed through monitoring of tumor metabolism using 18Fludeoxyglucose (FDG) PET-CT or 68Ga-PSMA-11 PET/CT for prostate cancer patients.
Exploratory outcomes: Immune monitoring of the tumor | 5 years
  Tumor immune profile will be assessed by multiplexed immunohistochemistry, tumor immunophenotyping, RNA expression as well as flow cytometry, ELISA and ELISPOT (enzyme-linked immunospot) assays.
Exploratory outcomes: Immune monitoring of the tumor microenvironment | 5 years
  Tumor microenvironment immune profile will be assessed by multiplexed immunohistochemistry, tumor immunophenotyping, RNA expression as well as flow cytometry, ELISA and ELISPOT (enzyme-linked immunospot) assays.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No